CLINICAL TRIAL: NCT02110394
Title: Observational Program for Evaluation of Ribomustin Use in the First Line Therapy of Chronic Lymphocytic Leukemia
Brief Title: Ribomustin in the First Line Therapy of Chronic Lymphocytic Leukemia
Acronym: NORMA
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: RU-BEN-NI-003
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: observational; chronic lymphocytic leukemia; bendamustine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bendamustine and rituximab
  Interventions: Other: bendamustine; Other: rituximab

INTERVENTIONS:
Other: bendamustine — Routine practice
  Other Names: Ribomustin
Other: rituximab — Routine practice
  Other Names: Mabthera

SUMMARY:
Prospective multicenter observational non-interventional study to assess routine clinical practice of Bendamustine use in the first line therapy of chronic lymphocytic leukemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic leukemia (CLL) with current or planned first line therapy with Ribomustin
* Informed Consent Form for personal data handling signed by the program participant

Exclusion Criteria:

* Any prior chemotherapy and/or radiotherapy and/or immunotherapy and/or any investigational agent for treatment of CLL
* Currently participating in any clinical trial, and/or has taken an investigational drug within 28 days prior to enrollment
* Contraindications for Ribomustin usage in accordance with product label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with В-cell chronic lymphocytic leukemia under the care of a physician in the haematology/chemotherapy departments in 20-25 centers in the Russian Federation
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Within 60-90 days after end of treatment

SECONDARY OUTCOMES:
Adverse drug reactions | At all post-treatment visits (up to 30 days after end of treatment)
Treatment Failure (TF) | Within 60-90 days after end of treatment
Time to Progression (TTP) | 60 months
Progression-Free Survival (PFS) | 60 months
Relapse following complete or partial remission | 60 months
Overall survival | 60 months
Quality of Life of patients receiving Ribomustin therapy | At all post-treatment visits (up to 30 days after end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (34):
- Russia (34):
  - Republic Clinical Hospital n.a. N.A. Semashko, Buryatia, Ulan-Ude
  - Alexandro-Mariinskaia Regional Clinical Hospital/13, Astrakhan
  - Vologda Reginal Clinical Hospital #2, Cherepovets
  - Irkutsk Regional Clinical Hospital/08, Irkutsk
  - Kaliningrad City Clinical Hospital, Kaliningrad
  - Regional Clinical Hospital#1/04, Khabarovsk
  - District Cancer Center od Khanty -Mansiysk, Khanty-Mansiysk
  - National Medical Surgical Center n.a.N.I.Pirogov/15, Moscow
  - RONC n.a.N.N.Blokhin/21, Moscow
  - Сentral Clinical Hospital n.a.N.A.Semashko/20, Moscow
  - Central Clinical Hospital of Department of Presidential Affairs, Moscow
  - Haematology Centre at Main Military Clinical Hospital n.a. N.N. Burdenko, Moscow
  - Murmansk Regional Clinical Hospital n.a.P.A.Bayandin/31, Murmansk
  - Nizhniy Novgorod Regional Clinical Hospital n.a.N.A.Semashko/14, Nizhny Novgorod
  - Medical Radiology Scientific Center/23, Obninsk
  - Omsk Regional Clinical Hospital, Omsk
  - Orenburg State Medical Academy/011, Orenburg
  - Perm regional hospital, Perm
  - Karelia Republican Сlinical Hospital n.a.V.A.Baranov/32, Petrozavodsk
  - Pskov Regional Clinical Hospital, Pskov
  - Rostov Scientific Research Oncology Institution/03, Rostov-on-Don
  - Site 70001 Private Practice, Saint Petersburg
  - Military-Medical Academy n.a. Kirova, Saint Petersburg
  - Samara State Medical University' Clinics/28, Samara
  - Saratov State Medical University n.a. V.I.Razumovskiy, Saratov
  - Road Clinical Hospital on Smolensk station OAO RZhD/12, Smolensk
  - Komi Republican Oncology Dispensary /01, Syktyvkar
  - Tula Regional Clinical Hospital/07, Tula
  - Tyumen Regional Clinical Hospital#1/27, Tyumen
  - Regional Clinical Hospital/26, Ulyanovsk
  - Volgograd Regional Clinical Oncology Dispensary#1/25, Volgograd
  - Vologda Regional Clinical Hospital, Vologda
  - Yekaterinburg City Hospital #7, Yekaterinburg
  - Yekaterinburg Regional Clinical Hospital #1, Yekaterinburg